CLINICAL TRIAL: NCT01519973
Title: Optimization of SPECT Cardiac Imaging Through Compensation for Attenuation, Resolution Loss and Scatter - The OSCARS
Brief Title: Optimization of SPECT Imaging
Acronym: OSCARS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment base changed due to change in clinical acquisition procedures
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Terrence Ruddy, Terrence Ruddy, MD, Ottawa Heart Institute Research Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HI Protocol #2008012-01H
Record Dates: First submitted 2011-07-15; First posted 2012-01-27 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Coronary Artery Disease
Keywords: Diagnostic imaging; Single Photon Emission Computed Tomography; Positron emission tomography; Computed tomography; Attenuation; Resolution; Scatter; Radiopharmaceutical
MeSH Terms: conditions — Coronary Artery Disease | interventions — Biological Evolution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Evaluation of technology in SPECT (Other): Evaluation of the accuracy of SPECT with new technologies for attenuation correction (AC), scatter correction (SC) and resolution recovery (RR) for assessment of myocardial perfusion using Rb-82 PET as the gold standard.
  Interventions: Radiation: SPECT/CT processed with Evolution for CardiacTM software

INTERVENTIONS:
Radiation: SPECT/CT processed with Evolution for CardiacTM software — SPECT/CT to be compared with PET/CT

SUMMARY:
Single Photon Emission Computed Tomography (SPECT) is a 3D nuclear medicine imaging technique that is used extensively to study the heart and diagnose heart disease. There are three major limitations in SPECT imaging: attenuation or loss of signal, scattering of the signal in the patient tissues and resolution, where the signal gets blurrier the further the nuclear activity is away from the camera. New software, Evolution for CardiacTM, by GE Healthcare and new cameras with computed tomography (CT) decrease the time needed for images to be obtained while maintaining image quality. Evaluation is needed before they become standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Intermediate to high risk patients with coronary artery disease who are scheduled for routine SPECT or PET perfusion imaging

Exclusion Criteria:

* Pregnancy and breast feeding
* Severe narrowing (stenosis) of the aortic valve
* Severe heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
• Determine the accuracy of myocardial perfusion assessment using SPECT with AC/SC/RR compared to Rb-82 PET. | 2 years
  We are proposing a study to evaluate the accuracy of SPECT with the new technologies for attenuation correction (AC), scatter compensation (SC) and resolution recovery (RR) for the assessment of myocardial perfusion in patients with heart disease using Rb-82 perfusion PET as the gold standard for comparison.

SECONDARY OUTCOMES:
Determine the incremental benefit of AC/SC/RR compared to AC alone | 2 years
Evaluate the effect on accuracy of using software with RR to reduce the acquisition time to half of the standard time. | 2 years
Determine if using a registered diagnostic CT (PET) increases the accuracy of CT-based AC over the lower-quality Hawkeye CT (SPECT). | 2 years
Determine if using a single CT scan acquired at stress for attenuation correction of both stress and rest SPECT decreases the accuracy over using CT scans acquired separately at rest and stress. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Terrence D Ruddy, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
This trial has concluded and the investigators have published from the available data.

REFERENCES:
- [Result] Wells RG, Soueidan K, Vanderwerf K, Ruddy TD. Comparing slow- versus high-speed CT for attenuation correction of cardiac SPECT perfusion studies. J Nucl Cardiol. 2012 Aug;19(4):719-26. doi: 10.1007/s12350-012-9555-4. Epub 2012 Apr 21. PMID 22527797
- [Result] Wells RG, Soueidan K, Timmins R, Ruddy TD. Comparison of attenuation, dual-energy-window, and model-based scatter correction of low-count SPECT to 82Rb PET/CT quantified myocardial perfusion scores. J Nucl Cardiol. 2013 Oct;20(5):785-96. doi: 10.1007/s12350-013-9738-7. Epub 2013 Jun 5. PMID 23737161